CLINICAL TRIAL: NCT04161768
Title: Comparative Study of Norfloxacin Versus Norfloxacin With Itopride in Secondary Prophylaxis of Spontaneous Bacterial Peritonitis
Brief Title: Norfloxacin With Itopride Versus Norfloxacin in Secondary Prophylaxis of Spontaneous Bacterial Peritonitis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SBP Management
Record Dates: First submitted 2019-11-10; First posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Spontaneous Bacterial Peritonitis
MeSH Terms: interventions — Norfloxacin; itopride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norfloxacin (Active Comparator): Norfloxacin 400 mg daily
  Interventions: Drug: Norfloxacin
- Norfloxacin and Itopride (Experimental): Norfloxacin 400 mg daily and Itopride 50 mg three times daily.
  Interventions: Drug: Norfloxacin; Drug: Itopride

INTERVENTIONS:
Drug: Norfloxacin — Norfloxacin 400 mg daily
  Other Names: Epinor
Drug: Itopride — Itopride 50 mg three times daily
  Other Names: Ganaton
  Arms: Norfloxacin and Itopride

SUMMARY:
Norfloxacin versus Norfloxacin with Itopride in Secondary Prophylaxis of Spontaneous Bacterial Peritonitis

DETAILED DESCRIPTION:
Comparative Study of Norfloxacin versus Norfloxacin with Itopride in Secondary Prophylaxis of Spontaneous Bacterial Peritonitis

ELIGIBILITY:
Inclusion Criteria:

* cirrhotic patients with ascites who had previous episodes of SBP.

Exclusion Criteria:

* 1. Allergy or contraindication for the used drugs. 2. Recent antibiotics therapy in the previous 2 weeks. 3. Patients with hepatocellular carcinoma or other neoplasia. 4. Pregnant and lactating women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of bouts of recurrence during treatment. | 6 months
  The recurrence of infection during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Afaf Younes Mohammed Younes, Msc, Principal Investigator — Tanta University - Faculty of Medicine; Mona Ahmed Helmy Shehata, Prof., Principal Investigator — Tanta University - Faculty of Medicine; Sherief Abd-Elsalam, Ass. Prof., Principal Investigator — Tanta University - Tropical Medicine Department
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No